CLINICAL TRIAL: NCT01700335
Title: Phase I Clinical Trial of SyB L-1101 in Patients With Myelodysplastic Syndrome
Brief Title: Safety and Pharmacokinetics Study of SyB L-1101 in Patients With Recurrent/Relapsed or Refractory Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011005
Record Dates: First submitted 2012-08-07; First posted 2012-10-04 (Estimated); Results first posted 2016-09-14 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- SyB L-1101 (Experimental): In Cohort 1, SyB L-1101 1200 mg/day group, Participants were administered 1200 mg/day of SyB L-1101 intravenously for 3 consecutive days, followed by 11-day observation period.
  In Cohort 2, SyB L-1101 1800 mg/day group, Participants were administered 1800 mg/day of SyB L-1101 intravenously for 3 consecutive days, followed by 11-day observation period.
  For both Cohorts, the treatment period of 14 days constitutes 1 cycle, and the treatment was allowed for up to 8 cycles.
  Interventions: Drug: SyB L-1101

INTERVENTIONS:
Drug: SyB L-1101 — SyB L-1101（rigosertib sodium） will be administered to two cohorts at either 1200 mg/day or 1800 mg/day.
  The dose will be administered intravenously for 72 continuous hours (3 days), followed by 11-day observation period. The treatment period of 14 days (3 days of administration + 11 days of observation) constitutes 1 cycle.
  The study will involve treatment through the second cycle, but treatment can be continued for 3 or more cycles if conditions for continued administration are satisfied.

SUMMARY:
The purpose of this study is to investigate tolerability when SyB L-1101 is administered intravenously in patients with recurrent/relapsed or refractory myelodysplastic syndrome, to determine the dose-limiting toxicity and maximum tolerated dose, and to estimate the recommended dose for phase II studies. Pharmacokinetics and antitumor effects will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

- Patients must satisfy the following conditions listed below.

1. Patients who have been histologically documented or cytologically confirmed with myelodysplastic syndrome (MDS), and who have been found to meet any of the following criteria on the basis of the World Health Organization (WHO) classification or French-American-British (FAB) classification.

   * Refractory Anemia (RA) (< 5% myeloblasts, < 15% ringed sideroblasts)
   * RA with Ring Sideroblasts (RARS) (< 5% myeloblasts, >= 15% ringed sideroblasts)
   * RA with Excess of Blasts (RAEB)-1 (5% to 9% myeloblasts)
   * RAEB-2 (10% to 19% myeloblasts)
   * RAEB in transformation (RAEB-t) (20% to 29% myeloblasts or < 25,000/mm^3 peripheral leukocytes)
   * Chronic myelomonocytic leukemia (CMML) (10% to 19% myeloblasts in marrow, >= 1,000/mm^3 peripheral monocytes, < 13,000/mm^3 leukocytes) However, RA patients must have score of Int-2 or higher in International prognostic scoring system (IPSS).
2. Patients with a low value in at least one blood cell lineage (having at least one of the following cytopenias).

   * Neutrophils : < 1,800/mm^3
   * Platelets : < 100,000/mm^3
   * Hemoglobin : < 10 g/dL
3. Patients with a previous history of chemotherapy (including lenalidomide) for the target disease who meet any of the following criteria.

   * Patients who have not achieved complete remission, partial remission, or hematologic improvement*
   * Patients with recurrence/relapse after complete remission, partial remission, or hematologic improvement*
   * Patients with intolerability that has led to discontinuation of treatment because of the development of liver dysfunction, kidney dysfunction, etc., after the start of treatment. * Proximate therapeutic efficacy judged under International Working Group (IWG) 2006 criteria
4. Patients who have not been treated for four weeks or longer after the end of the previous therapy and who are judged to have no residual effects (antitumor effects) from the previous therapy.
5. Patients who can be expected to survive at least three months or longer.
6. Patients at least 20 years old (when informed consent is obtained).
7. Patients who have score of 0 to 2 in Eastern Cooperative Oncology Group (ECOG) Performance Status (P.S.).
8. Patients with adequate function in major organs (heart, lungs, liver, kidneys, etc.).

   * Aspartate aminotransferase (AST) (Glutamic oxaloacetic transaminase, GOT) : no greater than 3.0 times the upper boundary of the reference range at each institution
   * Alanine aminotransferase (ALT) (Glutamic pyruvic transaminase, GPT): no greater than 3.0 times the upper boundary of the reference range at each institution
   * Total bilirubin: no more than 1.5 times the upper boundary of the reference range at each institution
   * Serum creatinine: no more than 1.5 times the upper boundary of the reference range at each institution
   * ECG: no abnormal findings requiring treatment
   * Echocardiography: no abnormal findings requiring treatment
9. Patients who personally signed an informed consent document for participation in this study.

Exclusion Criteria:

- Patients who satisfy any of the following conditions will not be enrolled in the study.

1. Patients with anemia caused by factors other than MDS (hemolytic anemia, gastrointestinal (GI) bleeding, etc.).
2. Patients who have undergone treatment for an active malignant tumor within the past year (except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast).
3. Patients who have been administered a cytokine preparation such as granulocyte-colony stimulating factor (G-CSF), erythropoietin, etc. within 14 days of tests for enrollment of the study.
4. Patients with obvious infectious diseases (including viral infections).
5. Patients with serious complications (liver failure, renal failure, etc.).
6. Patients with a complicating or previous history of serious heart disease (myocardial infarction, ischemic heart disease, etc.) within the past two years before enrollment, and with cardiac arrhythmia requiring treatment.
7. Patients with a serious gastrointestinal condition (severe or significant nausea/vomiting, diarrhea, etc.).
8. Patients who are positive for the Hepatitis B surface (HBs) antigen or HIV antibodies.
9. Patients with serious bleeding tendencies (disseminated intravascular coagulation (DIC), internal hemorrhage, etc.).
10. Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 mEq/L).
11. Patients who have been administered a drug in a clinical trial or an unapproved drug within three months before enrollment.
12. Patients with an addiction to a legal or illegal drug, or with alcohol dependency.
13. Patients who are pregnant or may become pregnant.
14. Patients who have not consented to the following contraceptive measures.

    Patients will avoid sexual intercourse with sexual partners or should use the following contraceptive methods in these time periods: for male patients during the administration period of the trial and for six months after the end of administration; female patients during the administration period of the trial, and until a second menstrual period is confirmed after the end of administration (or in the case of female patients with no menstrual period, for two months after the end of administration).

    •Male patients

    The patient will always use a condom. For effective contraception, it is recommended that the female partner also use the contraceptive methods for female patients.

    •Female patients

    Female patients who may become pregnant should use one or more types of the following contraceptive methods. In addition, the male partner will always use a condom.
    * Oral contraceptive (birth control pills)
    * Intrauterine device (IUD)
    * Tubal ligation
15. Other patients judged to be unsuitable by an investigator or sub-investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukuoka
  - Research Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- SyB L-1101 1200 mg/Day Group: Cohort 1: Participants were administered 1200 mg/day of SyB L-1101 intravenously for 3 consecutive days, followed by 11-day observation period.
  The treatment period of 14 days constitutes 1 cycle, and the treatment was allowed for up to 8 cycles.
- SyB L-1101 1800 mg/Day Group: Cohort 2: Participants were administered 1800 mg/day of SyB L-1101 intravenously for 3 consecutive days, followed by 11-day observation period.
  The treatment period of 14 days constitutes 1 cycle, and the treatment was allowed for up to 8 cycles.
Period: Overall Study
Arm/Group | SyB L-1101 1200 mg/Day Group | SyB L-1101 1800 mg/Day Group
Started | 3 | 6
Completed | 2 | 2
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received at least 1 dose of SyB L-1101 either at 1200 mg/day or 1800 mg/day intravenously.
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Customized [Number; unit: participants]
  60-69 years | 4
  70-79 years | 4
  80- years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as adverse events for which a causal relationship with the investigational drug could not be ruled out and which met the following criteria that occurred by the final observation in Cycle 2. DLTs were also to be assessed in the Efficacy and Safety Assessment Committee.
  Criteria:
  1. Grade 3 or higher non-hematologic toxicity. However, nausea, vomiting, diarrhea, pyrexia, stomatitis, and esophagitis/dysphagia are excluded (Grade 3 nausea, vomiting, diarrhea, and pyrexia that cannot be controlled with antiemetic, antidiarrheal, or antifebrile agents are regarded as DLTs)
  2. Grade 3 or higher stomatitis, esophagitis, and dysphagia that persist for >= 4 days
Time Frame: Up to 60 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101 1200 mg/Day Group | SyB L-1101 1800 mg/Day Group
Number analyzed (Participants) | 3 | 6
participants | 0 | 2

2. Secondary Outcome: Hematologic Remission Effect (IWG 2006 Criteria, Responses Must be Sustained at Least 4 Weeks)
Description: Definition
  Complete remission (CR) Bone marrow: <= 5% myeloblasts; normal maturation of all cell lines Peripheral blood: Hemoglobin (Hgb) >= 11 g/dL, Platelets >= 100×10^9/L, Neutrophils >= 1.0×10^9/L, Blasts 0%
  Partial remission (PR) Same as CR criteria except bone marrow blasts decreased by >= 50% over pretreatment but still > 5%
  Marrow CR Bone marrow: <= 5% myeloblasts and decrease by >= 50% over pretreatment Peripheral blood: will be noted in addition to marrow CR
  Stable disease Failure to achieve at least PR, but no evidence of progression for > 8 wks
  Disease progression
  Patients with:
  Less than 5% blasts: >= 50% increase in blasts to > 5% blasts 5%-10% blasts: >= 50% increase to > 10% blasts 10%-20% blasts: >= 50% increase to > 20% blasts 20%-30% blasts: >= 50% increase to > 30% blasts
  Any of the following:
  At least 50% decrement from maximum remission/response in granulocytes or platelets Reduction in Hgb by >= 2 g/dL Transfusion dependence
Time Frame: Up to 60 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101 1200 mg/Day Group | SyB L-1101 1800 mg/Day Group
Number analyzed (Participants) | 3 | 6
participants
  CR | 0 | 0
  PR | 0 | 0
  Marrow CR | 0 | 0
  Stable disease (SD) | 0 | 2
  Treatment failure | 0 | 0
  Disease progression | 3 | 2
  Not assessable | 0 | 2
  Remission rate | 0 | 0

3. Secondary Outcome: Hematologic Improvement Effect (IWG 2006 Criteria, Responses Must be Sustained at Least 8 Weeks)
Description: Definition
  Hematologic Improvement Erythrocyte (HI-E):
  Hgb increase by >= 1.5 g/dL Relevant reduction of units of red blood cell (RBC) transfusions by an absolute number of at least 4 RBC transfusions/8 week compared with the pretreatment transfusion number in the previous 8 week. Only RBC transfusions given for a Hgb of <= 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation
  Hematologic Improvement Platelet (HI-P):
  Absolute increase of >= 30×10^9/L for patients starting with > 20×10^9/L platelets Increase from < 20×10^9/L to > 20×10^9/L and by at least 100%
  Hematologic Improvement Neutrophil (HI-N):
  At least 100% increase and an absolute increase > 0.5×10^9/L
  Progressive disease / Relapse:
  At least 1 of the following:
  At least 50% decrement from maximum response levels in granulocytes or platelets Reduction in Hgb by >= 1.5 g/dL Transfusion dependence
Time Frame: Up to 60 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101 1200 mg/Day Group | SyB L-1101 1800 mg/Day Group
Number analyzed (Participants) | 3 | 6
participants
  HI-E | 0 | 0
  HI-P | 0 | 0
  HI-N | 0 | 0
  Progressive disease | 1 | 2
  Relapse | 0 | 0
  Not assessable | 2 | 4
  Hematologic improvement rate | 0 | 0

4. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was investigated with an index of DLT
Time Frame: Up to 16 weeks
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 9
participants | NA — MTD was not reached

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | SyB L-1101 1200 mg/Day Group | SyB L-1101 1800 mg/Day Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB L-1101 1200 mg/Day Group (N=3) | SyB L-1101 1800 mg/Day Group (N=6)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB L-1101 1200 mg/Day Group (N=3) | SyB L-1101 1800 mg/Day Group (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (1)
Tongue haematoma (Gastrointestinal disorders) | 1 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (3)
Oedema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (4)
Thirst (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 1 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (2)
Lymphocyte count decreased (Investigations) | 2 (6) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (6) | 2 (3)
Platelet count decreased (Investigations) | 2 (3) | 4 (6)
Protein total decreased (Investigations) | 1 (1) | 1 (2)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (3)
White blood cell count decreased (Investigations) | 2 (3) | 3 (9)
Neutrophil percentage decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte percentage increased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2)
Hepatitis B DNA assay positive (Investigations) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 3 (6)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No